CLINICAL TRIAL: NCT02010047
Title: A Study to Compare the Performance of a qPCR-based Assay to Immunohistochemistry (IHC) and Fluorescence in Situ Hybridization (FISH) in the Detection of Anaplastic Lymphoma Kinase (ALK) Fusion Mutations in Formalin Fixed Paraffin-embedded (FFPE) Tissue From Non-small Cell Lung Cancer (NSCLC) Patients.
Brief Title: Comparison of qPCR to IHC and FISH for Detection of ALK Fusion Mutations in FFPE Tissue From NSCLC Patients
Acronym: PCRTALK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Insight Genetics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PCRTALK
Record Dates: First submitted 2013-12-05; First posted 2013-12-12 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2014-07

CONDITIONS: Nonsmall Cell Lung Cancer
Keywords: Anaplastic lymphoma kinase gene; Polymerase chain reaction; Immunohistochemistry; Fluorescence in situ hybridization
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IHC, FISH and qPCR ALK assays (Experimental): ALK testing by IHC and FISH will be compared to ALK qPCR testing on NSCLC FFPE tissue.
  Interventions: Device: ALK qPCR assay

INTERVENTIONS:
Device: ALK qPCR assay — 72 IHC ALK-negative and 72 IHC ALK-positive FFPE samples will tested with FISH and qPCR to determine the sensitivity and specificity of the ALK qPCR assay.

SUMMARY:
The anaplastic lymphoma kinase gene(ALK) is mutated approximately 5% of non-small cell lung cancers. Testing for this gene is important because there are drugs known as ALK inhibitors that have been shown to significantly delay the progression of ALK-mutated lung cancers. There are a number of ways to test for the presence of the ALK gene in lung cancer biopsy tissue. One method involves making slides and staining them to detect the ALK protein. This is called immunohistochemistry. Another method called fluorescence in situ hybridization(FISH)is used to detect rearrangements of the ALK gene associated with lung cancer. Although both these tests are widely used to test for ALK gene abnormalities, the techniques may not always find the ALK gene mutation because they are not sensitive enough or not enough cancer cells are present in the lung biopsy.

This study is being performed to determine if a technique called quantitation polymerase chain reaction (qPCR) is as accurate or better at finding the ALK gene mutation in lung cancer biopsy tissue.

ELIGIBILITY:
Inclusion Criteria:

* You have a confirmed diagnosis of non-squamous, non-endocrine non-small cell lung cancer.
* Your cancer biopsy has sufficient cancer cells to be tested for the (Epidermal Growth Factor Receptor (EGFR) mutation, the ALK fusion gene abnormality and the research ALK testing.
* Your lung cancer biopsy is determined not to have a mutation in the EGFR gene.
* You are 19 years old or older.
* You fully understand the study and give informed consent to participate as demonstrated by signing the consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08-18 (Actual); Study Completion 2015-08-18 (Actual)

PRIMARY OUTCOMES:
To determine the true number of ALK positives and negatives of a qPCR assay for the detection in FFPE lung cancer biopsy specimens of ALK status in comparison with IHC and FISH ALK detection technologies. | Up to 24 weeks after the completing of enrollment of 72 ALK negative and 72 ALK positive tumor blocks

SECONDARY OUTCOMES:
The analysis of plasma and serum collected from those patients with ALK-positive NSCLC to assess the feasibility for the use of non-invasive sampling in the diagnosis and disease monitoring of lung cancer. | After completion of enrollemnt of 72 ALK postive tumor blocks.

CONTACTS AND LOCATIONS:
Overall Officials: David L Saltman, MD PhD, Principal Investigator — British Columbia Cancer Agency; Aly Karsan, MD, Principal Investigator — BC Cancer Agency, Molecular Diagnostic Laboraotry
Locations (7):
- Canada (7):
  - BC Cancer Agency-Abbotsford Centre, Abbotsford, British Columbia
  - BC Cancer Agency-Centre for the Southern Interior, Kelowna, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - BC Cancer Agency-Centre for the North, Prince George, British Columbia
  - BC Cancer Agency, Frase Valley Centre, Surrey, British Columbia
  - BC Cancer Agency, Vancouver Centre, Vancouver, British Columbia
  - BC Cancer Agency, Victoria, British Columbia